CLINICAL TRIAL: NCT05035186
Title: Efficacy of Clarithromycin and Flouroquinolones Based Regimens in H.Pylori Eradication in Covid-19 Era: a Randomized Controlled Trial
Brief Title: Efficacy of Clarithromycin and Flouroquinolones Based Regimens in H.Pylori Eradication in Covid-19 Era
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Kamal, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0305083
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Levofloxacin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Clarithromycin based
  Interventions: Drug: Amoxicillin
- Group 2 (Experimental): Levofloxacin based
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — Anti-H. pylori regimens
  Other Names: Clarithromycin; Levofloxacin

SUMMARY:
Era of COVID-19 and the related panic lead to widely spread antibiotics misuse especially for azithromycin. Cross sensitivity between azithromycin and clarithromycin can impact success rates of H. pylori treatment regimens.(1) Here we aim to explore this point in Egyptian patients.

Sample size Supposing the cure rate of clarithromycin-based regimen to levofloxacin based regimen is 69% versus 84.5% respectively. Using Medcalc, the minimal required sample size is 116 patients for each arm (type 1 error= 5%, type II error=20%). Each arm increased by 10% to compensate for drop-out. The sample size will be 135 for each arm.

Study Arms:

* Arm 1: The first group will receive (amoxicillin 1g/12 hrs, Clarithromycin 500 mg/12hrs, esomeprazole 40mg/12hrs)
* Arm 2: The second group will receive (esomeprazole 40 mg/12hrs, levofloxacin 500 mg/24 hrs, and amoxicillin 1gm/12 hrs).
* To confirm patient compliance, we will ask patients to bring their remaining medication and counted the rest of their pills. Patients with a compliance of <80% will be excluded from the study per protocol (PP) analysis.

ELIGIBILITY:
Inclusion Criteria:

* • Patients aged 18-65 years old with newly diagnosed positive H. pylori antigen in stools, urea breath test or H. pylori detected on endoscopy.

Exclusion Criteria:

* • Women who are pregnant or lactating, patients previously treated with H. pylori eradication therapy, those with recent exposure to antibiotics within the previous 3 months, patients who previously underwent gastric surgery, patients with malignant neoplasms, and patients with other severe concomitant diseases like renal, hepatic impairement, heart failure NYHA class II or more, hypoalbuminemia and those with possible clinically significant drug-drug interaction with any of the study's drugs will be excluded.

  * Known allergy to antibiotics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rates | 6 weeks from end of treatment and at least 2 weeks with no administration of PPIs

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kamal, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University., Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kamal A, Ghazy RM, Sherief D, Ismail A, Ellakany WI. Helicobacter pylori eradication rates using clarithromycin and levofloxacin-based regimens in patients with previous COVID-19 treatment: a randomized clinical trial. BMC Infect Dis. 2023 Jan 20;23(1):36. doi: 10.1186/s12879-023-07993-8. PMID 36670359